CLINICAL TRIAL: NCT03099187
Title: Multicenter, International, Double-blind, Two-Arm, Randomized, Placebo-controlled Phase II Trial of Pirfenidone in Patients With Unclassifiable Progressive Fibrosing ILD
Brief Title: A Study of Pirfenidone in Patients With Unclassifiable Progressive Fibrosing Interstitial Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA39189; 2016-002744-17 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-04 (Actual); Results first posted 2020-01-03 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pirfenidone (Experimental): Participants will receive pirfenidone 267 mg capsule three times a day from Day 1 to 7 followed by 2 capsules three times a day from Day 8 to 14 then 3 capsules three times a day from Day 15 up to Week 24.
  Interventions: Drug: Pirfenidone
- Placebo (Experimental): Participants will receive matching placebo capsule three times a day from Day 1 to 7 followed by 2 capsules three times a day from Day 8 to 14 then 3 capsules three times a day from Day 15 up to Week 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone 267 mg capsules three times in a day.
  Arms: Pirfenidone
Drug: Placebo — Matching placebo capsules three times in a day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pirfenidone in participants with fibrosing interstitial lung disease (ILD) who cannot be classified with moderate or high confidence into any other category of fibrosing ILD by multidisciplinary team (MDT) review ("unclassifiable" ILD).

DETAILED DESCRIPTION:
Study participants will be randomised to receive 801 mg pirfenidone or placebo three times daily for 24 weeks. The efficacy of pirfenidone versus placebo will be assessed by daily measurement of forced vital capacity using a handheld spirometer over the treatment period. Additionally, the study will assess the efficacy and safety of pirfenidone with and without concomitant mycophenolate mofetil treatment and in study participants with or without interstitial pneumonia with autoimmune features (IPAF). All study participants who attend the follow-up visit at Week 28 will be offered the opportunity to receive open-label pirfenidone within the trial protocol. In order to maintain blinding of the controlled period of the study, all study participants will discontinue treatment by Week 24 and return for a follow-up visit 4 weeks later. Study participants eligible to participate in the single-arm 12-month extension will be initiated on open-label pirfenidone during this visit (re-starting the dose titration from one capsule three times daily [TID]). During the long-term extension period, study participants will be monitored for safety, initially at monthly visits during the first 6 months and thereafter approximately every 3 months. A final follow-up visit will take place 4 weeks after the last dose of pirfenidone is taken.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18-85 years
* Confirmed fibrosing ILD which, following multidisciplinary team review, cannot be classified with either high or moderate confidence as a specific idiopathic interstitial pneumonia or other defined ILD
* Progressive disease as considered by the investigator as participants deterioration within the last 6 months, which is defined as a rate of decline in forced vital capacity (FVC) >5% or a significant symptomatic worsening not due to cardiac, pulmonary vascular or other causes
* Extent of fibrosis >10% on high-resolution computed tomography
* Forced vital capacity >= 45% of predicted value
* Diffusing capacity of the lung for carbon monoxide (DLco) >= 30% of predicted value
* Forced expiratory volume in 1 second/FVC ratio >= 0.7
* Able to do 6-minute walk distance (6MWD) >= 150 meters
* For women of childbearing potential: agreement to remain abstinent or use a non-hormonal or hormonal contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of pirfenidone
* For men, agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Diagnosis with moderate or high confidence of nonspecific interstitial pneumonia and any ILD with an identifiable cause such as connective tissue disease-ILD, chronic hypersensitivity pneumonitis, or others
* Diagnosis of idiopathic pulmonary fibrosis independent of the confidence level
* History of unstable angina or myocardial infarction during the previous 6 months
* Treatment with high dose systemic corticosteroids, or any immunosuppressant other than mycophenolate mofetil/acid (MMF), at any time within the 4 weeks of the screening period. Participants being treated with MMF should be on a stable dose that is expected to remain stable throughout the trial and was started at least 3 months prior to screening
* Participants previously treated with pirfenidone or nintedanib
* Participants treated with N-acetyl-cysteine for fibrotic lung disease, at any time within the 4 weeks of the screening period
* Drug treatment for any type of pulmonary hypertension
* Participation in a trial of an investigational medicinal product within the last 4 weeks
* Significant other organ co-morbidity including hepatic or renal impairment
* Predicted life expectancy < 12 months or on an active transplant waiting list
* Use of any tobacco product in the 12 weeks prior to the start of screening, or any unwillingness to abstain from their use through to the Follow-up Visit
* Illicit drug or alcohol abuse within 12 months prior to screening
* Planned major surgery during the trial
* Hypersensitivity to the active substance or to any of the excipients of pirfenidone
* History of angioedema
* Concomitant use of fluvoxamine
* Clinical evidence of any active infection
* Any history of hepatic impairment, elevation of transaminase enzymes, or liver function test results as: Total bilirubin above the upper limit of normal (ULN), Aspartate aminotransferase or alanine aminotransferase >1.5 × ULN, and Alkaline phosphatase >2.0 × ULN
* Creatinine clearance < 30 milliliter (mL) per minute, calculated using the Cockcroft-Gault formula
* Any serious medical condition, clinically significant abnormality on an Electrocardiogram (ECG) at screening, or laboratory test results
* An ECG with a heart rate corrected QT interval using Fridericia's formula as >= 500 milliseconds at screening, or a family or personal history of long QT syndrome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (66):
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - John Hunter Hospital; Respiratory Department; Respiratory Department, New Lambton Heights, New South Wales
  - Lung Research Queensland, Nundah, Queensland
  - Princess Alexandra Hospital, Department of Respiratory and Sleep Medicine, Woolloongabba, Queensland
  - Royal Adelaide Hospital; Respiratory Clinical Trials Unit, Thoracic Medicine, Adelaide, South Australia
  - Respiratory Department, Heidelberg, Victoria
  - The Alfred Hospital, Prahan, Victoria
  - Fiona Stanley Hospital; Advanced Lung Disease Unit, Murdoch, Western Australia
- Belgium (3):
  - ULB Hôpital Erasme, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Canada (2):
  - Pacifica Lung Research Center/St. Paul's Hospital, Vancouver, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
- Czechia (4):
  - Fakultni Nemocnice Brno-Bohunice; Klinika Tuberkulozy A Respiracnich Chorob, Brno
  - Nemocnice Jihlava, Jihlava
  - Fakultni nemocnice Olomouc; Pneumologicka klinika, Olomouc
  - Vseobecna fakultni nemocnice v Praze; I. klinika tuberkulozy a respiracnich nemoci, Prague
- Denmark (3):
  - Aarhus Universitetshospital; Lungesygdomme, Forskning, Aarhus N
  - Gentofte Hospital, Lungemedicinsk Afdeling, Hellerup
  - Odense Universitetshospital, Lungemedicinsk Afdeling J, Odense C
- Germany (5):
  - Zentralklinik Bad Berka GmbH; Pneumologie, Bad Berka
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Klinik der Justus-Liebig-Universität; Innere Medizin, Giessen
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Klinikum der Universität München; Campus Großhadern; Med. Klinik und Poliklinik V, München
- Greece (3):
  - Sotiria Hospital for Diseases of the Chest, Academic Department of Pneumonology, Athens
  - University General Hospital of Athens "Attikon", B' University Pulmonary Clinic, Chaïdári
  - University General Hospital of Heraklio, Pulmonary Clinic, Heraklio
- Ireland (2):
  - Mater Misericordiae University hospital, Dublin
  - St Vincents University Hospital, Dublin
- Israel (7):
  - Soroka; Pulmonary Clinic, Beersheba
  - Carmel Medical Center; Pulmonary Institute, Haifa
  - Shaare Zedek Medical Center; Pulmonary Inst., Jerusalem
  - Hadassah Medical Center; Pulmonary Institute, Jerusalem
  - Meir Medical Center; Pulmonary Dept, Kfar Saba
  - Beilinson Medical Center; Pulmonary Inst., Petah Tikva
  - Kaplan Medical Center, Rehovot
- Italy (5):
  - Ospedale Morgagni-Pierantoni; U.O. Pneumologia, Forlì, Emilia-Romagna
  - Ospedale San Giuseppe; U.O. di Pneumologia, Milan, Lombardy
  - A.O. Universitaria San Luigi Gonzaga di Orbassano; Ambulatorio per le Malattie Rare del Polmone, Orbassano (TO), Piedmont
  - A.O.U. Ospedali Riuniti Umberto I -G.M. Lancisi-G. Salesi Ancona; SOD Pneumologia, Torrette Di Ancona, The Marches
  - Azienda Ospedaliero-Universitaria Careggi; SOD Pneumologia e Fisiopatologia Toracico Polmonare, Florence, Tuscany
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne;Klinika Alergologii i Pneumonologii, Gdansk
  - Uniwersytecki Szpital Kliniczny Nr 1 im.N.Barlickiego Oddzial Kliniczny Pneumonologii i Alergologii, Lodz
  - Instytut Gruźlicy i Chorób Płuc, I Klinika Chorób Płuc, Warsaw
- Portugal (4):
  - Hospital Infante D. Pedro; Servico de Pneumologia, Aveiro
  - HUC; Servico de Pneumologia A, Coimbra
  - Hospital de Sao Joao; Servico de Pneumologia, Porto
  - CHVNG/E_Unidade 1; Servico de Pneumologia, Vila Nova de Gaia
- Spain (5):
  - Hospital Universitari de Bellvitge ; Servicio de Neumologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de neumologia, Santander, Cantabria
  - Hospital Universitario La Princesa; Servicio de Neumologia, Madrid
  - Hospital Clínico San Carlos - Servicio de Neumologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Neumologia, Madrid
- United Kingdom (12):
  - University Hospital Birmingham Queen Elizabeth Hospital, Birmingham
  - Southmead Hospital; Respiratory Department, Bristol
  - Papworth Hospital NHS Foundation Trust; Respiratory Department, Cambridge
  - Edinburgh Royal Infirmary; Respiratory Department, Edinburgh
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Glenfield Hospital, Leicester
  - University College London Hospital; Respiratory Medicine, London
  - Royal Brompton Hospital; Respiratory Department, London
  - Wythenshawe Hospital; North West Lung Research Centre, Manchester
  - Northern General Hospital, Sheffield
  - Southampton University Hospitals NHS Trust, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Molina-Molina M, Kreuter M, Cottin V, Corte TJ, Gilberg F, Kirchgaessler KU, Axmann J, Maher TM. Efficacy of Pirfenidone vs. Placebo in Unclassifiable Interstitial Lung Disease, by Surgical Lung Biopsy Status: Data From a post-hoc Analysis. Front Med (Lausanne). 2022 Jun 17;9:897102. doi: 10.3389/fmed.2022.897102. eCollection 2022. PMID 35783648
- [Derived] Kreuter M, Maher TM, Corte TJ, Molina-Molina M, Axmann J, Gilberg F, Kirchgaessler KU, Cottin V. Pirfenidone in Unclassifiable Interstitial Lung Disease: A Subgroup Analysis by Concomitant Mycophenolate Mofetil and/or Previous Corticosteroid Use. Adv Ther. 2022 Feb;39(2):1081-1095. doi: 10.1007/s12325-021-02009-w. Epub 2021 Dec 22. PMID 34936057
- [Derived] Maher TM, Corte TJ, Fischer A, Kreuter M, Lederer DJ, Molina-Molina M, Axmann J, Kirchgaessler KU, Samara K, Gilberg F, Cottin V. Pirfenidone in patients with unclassifiable progressive fibrosing interstitial lung disease: a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Respir Med. 2020 Feb;8(2):147-157. doi: 10.1016/S2213-2600(19)30341-8. Epub 2019 Sep 29. PMID 31578169
- [Derived] Graney BA, Fischer A. Interstitial Pneumonia with Autoimmune Features. Ann Am Thorac Soc. 2019 May;16(5):525-533. doi: 10.1513/AnnalsATS.201808-565CME. PMID 30695649
- [Derived] Maher TM, Corte TJ, Fischer A, Kreuter M, Lederer DJ, Molina-Molina M, Axmann J, Kirchgaessler KU, Cottin V. Pirfenidone in patients with unclassifiable progressive fibrosing interstitial lung disease: design of a double-blind, randomised, placebo-controlled phase II trial. BMJ Open Respir Res. 2018 Sep 4;5(1):e000289. doi: 10.1136/bmjresp-2018-000289. eCollection 2018. PMID 30233802

RESULTS

PARTICIPANT FLOW:
Groups:
- Pirfenidone: Participants received pirfenidone 267 mg capsule three times a day from Day 1 to 7 followed by 2 capsules three times a day from Day 8 to 14 then 3 capsules three times a day from Day 15 up to Week 24.
- Placebo: Participants received matching placebo capsule three times a day from Day 1 to 7 followed by 2 capsules three times a day from Day 8 to 14 then 3 capsules three times a day from Day 15 up to Week 24.
- Open-Label Treatment (Pirfenidone); Open-Label Treatment (Placebo): After participants completed the double-blind treatment period and the follow-up visit at Week 28, they were offered the option to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. A final follow-up visit was performed at the end of the safety period, 28 days after the last open-label dose.
Period: Double-blind Treatment
Arm/Group | Pirfenidone | Placebo | Open-Label Treatment (Pirfenidone) | Open-Label Treatment (Placebo)
Started | 127 | 126 | 0 | 0
Completed | 94 | 110 | 0 | 0
Not Completed | 33 | 16 | 0 | 0
Not completed — Adverse Event | 19 | 1 | 0 | 0
Not completed — Death | 1 | 3 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 4 | 0 | 0
Not completed — Lung transplantation | 0 | 1 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 2 | 0 | 0
Not completed — Disease progression | 0 | 1 | 0 | 0
Not completed — Randomization error | 0 | 2 | 0 | 0
Not completed — Non-compliance with Protocol procedure | 1 | 1 | 0 | 0
Period: 12-month Safety Follow-up
Arm/Group | Pirfenidone | Placebo | Open-Label Treatment (Pirfenidone) | Open-Label Treatment (Placebo)
Started | 0 | 0 | 94 | 110
Completed | 0 | 0 | 75 | 84
Not Completed | 0 | 0 | 19 | 26
Not completed — Adverse Event | 0 | 0 | 5 | 12
Not completed — Death | 0 | 0 | 7 | 9
Not completed — Lung transplantation | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Symptomatic deterioration | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 2
Not completed — Due to hospitalization | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pirfenidone: Participants received pirfenidone 267 mg capsule three times a day from Day 1 to 7 followed by 2 capsules three times a day from Day 8 to 14 then 3 capsules three times a day from Day 15 up to Week 24. After participants completed the double-blind treatment period and the follow-up visit at Week 28, they were offered the option to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. A final follow-up visit was performed at the end of the safety period, 28 days after the last open-label dose.
- Placebo: Participants received matching placebo capsule three times a day from Day 1 to 7 followed by 2 capsules three times a day from Day 8 to 14 then 3 capsules three times a day from Day 15 up to Week 24. After participants completed the double-blind treatment period and the follow-up visit at Week 28, they were offered the option to receive open-label pirfenidone within the trial protocol in a safety follow-up period of up to 12 months. A final follow-up visit was performed at the end of the safety period, 28 days after the last open-label dose.
- Total: Total of all reporting groups
Arm/Group | Pirfenidone | Placebo | Total
Number analyzed (Participants) | 127 | 126 | 253
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (10.1) | 67.7 (9.2) | 67.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114
  Male | 70 | 69 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 115 | 112 | 227
  Not reported | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian | 5 | 0 | 5
  Black or African American | 1 | 2 | 3
  Other | 0 | 1 | 1
  White | 120 | 123 | 243

OUTCOME MEASURES:

1. Primary Outcome: Rate of Decline in Forced Vital Capacity (FVC) Over the 24-week Double-blind Treatment Period
Description: Rate of decline in FVC was measured in mL by daily handheld spirometer. The analyses were repeated due to an additional independent review of the home spirometry data.
Time Frame: Up to Week 24
Population: The intent-to-treat (ITT) population was defined as all randomized participants. The ITT population was the primary analysis population for all efficacy analyses. Only participants for whom data were collected are included in the analysis.
Measure: Mean (95% Confidence Interval); unit: milliliter (mL)
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
milliliter (mL)
  Primary Analysis in 2019: number analyzed (Participants) | 124 | 123
  Primary Analysis in 2019 | -17.9 [-311.7 to 275.9] | 116.6 [-451.9 to 685.2]
  Final Analysis in 2020: number analyzed (Participants) | 116 | 116
  Final Analysis in 2020 | -90.3 [-157.0 to -23.7] | 125.6 [-458.4 to 709.6]
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019. Mean FVC decline comparison between treatment groups using a Student's t-test with a two-sided significance level of 0.05; Test type: Superiority; p = 0.6777, t-test, 2 sided — p-value was not adjusted for multiplicity and is provided for descriptive purpose only; Difference in Group Means = -134.6, 95% CI 2-sided [-772.4 to 503.3]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020. Mean FVC decline comparison between treatment groups using a Student's t-test with a two-sided significance level of 0.05; Test type: Superiority; p = 0.4682, Student's t-test — p-value was not adjusted for multiplicity and is provided for descriptive purpose only; Difference in Group Means = -216.0, 95% CI 2-sided [-803.6 to 371.7]

2. Secondary Outcome: Change in Percent Predicted FVC
Description: FVC was measured in liter (L) by spirometry. The analyses were repeated due to additional data cleaning activities that were not conducted during the primary analysis.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent predicted (%)
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Percent predicted (%)
  Baseline (Day 1) | 73.95 (18.815) | 73.95 (19.974)
  Week 4: number analyzed (Participants) | 120 | 121
  Week 4 | 74.04 (19.009) | 74.55 (21.223)
  Week 8: number analyzed (Participants) | 115 | 117
  Week 8 | 73.98 (19.324) | 73.50 (20.168)
  Week 12: number analyzed (Participants) | 110 | 114
  Week 12 | 73.96 (19.493) | 73.91 (20.856)
  Week 16: number analyzed (Participants) | 103 | 113
  Week 16 | 74.56 (20.299) | 72.65 (22.479)
  Week 20: number analyzed (Participants) | 102 | 115
  Week 20 | 73.94 (21.000) | 71.99 (21.673)
  Week 24: number analyzed (Participants) | 101 | 112
  Week 24 | 72.95 (20.819) | 73.55 (22.383)
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.0383, rank ANCOVA
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.0239, rank ANCOVA

3. Secondary Outcome: Change in FVC
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Liter (L)
  Baseline | 2.36 (0.793) | 2.38 (0.747)
  Week 4: number analyzed (Participants) | 120 | 121
  Week 4 | 2.37 (0.818) | 2.37 (0.786)
  Week 8: number analyzed (Participants) | 115 | 117
  Week 8 | 2.37 (0.822) | 2.36 (0.816)
  Week 12: number analyzed (Participants) | 110 | 114
  Week 12 | 2.37 (0.820) | 2.35 (0.773)
  Week 16: number analyzed (Participants) | 103 | 113
  Week 16 | 2.41 (0.860) | 2.31 (0.782)
  Week 20: number analyzed (Participants) | 102 | 115
  Week 20 | 2.40 (0.866) | 2.30 (0.796)
  Week 24: number analyzed (Participants) | 101 | 112
  Week 24 | 2.37 (0.863) | 2.34 (0.773)
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.0018, Student's t-test — p-value was not adjusted for multiplicity and was provided for descriptive purpose only; Overall Mean Difference = 95.3, 95% CI 2-sided [35.9 to 154.6]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.0096, Student's t-test — p-value was not adjusted for multiplicity and was provided for descriptive purpose only; Overall Mean Difference = 84.3, 95% CI 2-sided [20.7 to 147.8]

4. Secondary Outcome: Categorical Change in FVC of >5%
Description: Categorical change in FVC was measured both by daily spirometry as well as by spirometry during clinical visits. Only the site spirometry data were used as the daily spirometry data were not normally distributed. The analyses were repeated due to additional data cleaning activities that were not conducted during the primary analysis.
Time Frame: Baseline (Day 1) to Week 24
Population: The intent-to-treat (ITT) population was defined as all randomized participants. The ITT population was the primary analysis population for all efficacy analyses.
Measure: Number; unit: Number of Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Number of Participants
  Primary Analysis in 2019 | 47 | 74
  Final Analysis in 2020 | 47 | 73
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel — p-value was not adjusted for multiplicity and was provided for descriptive purpose only; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.25 to 0.69]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel — p-value was not adjusted for multiplicity and was provided for descriptive purpose only; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.26 to 0.71]

5. Secondary Outcome: Categorical Change in FVC of >10%
Description: as for outcome 4
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 4
Measure: Number; unit: Number of Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Number of Participants
  Primary Analysis in 2019 | 18 | 34
  Final Analysis in 2020 | 18 | 33
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.0114, Cochran-Mantel-Haenszel — p-value was not adjusted for multiplicity and was provided for descriptive purpose only; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.23 to 0.84]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.0168, Cochran-Mantel-Haenszel — p-value was not adjusted for multiplicity and was provided for descriptive purpose only; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.24 to 0.88]

6. Secondary Outcome: Change in Percent Predicted Diffusing Capacity of the Lung for Carbon Monoxide (DLco)
Description: The DLco is a pulmonary function test that measures the capacity for the lung to carry out gas exchange between the inhaled breath and the pulmonary capillary blood vessels and the DLco %-predicted represents the DLco expressed as a percentage of the expected normal valued based on the participant's age, height, gender and ethnicity.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
% predicted
  Baseline (Day 1): number analyzed (Participants) | 126 | 125
  Baseline (Day 1) | 46.19 (12.403) | 49.57 (13.931)
  Change from Baseline at Week 12 (Primary Analysis in 2019): number analyzed (Participants) | 110 | 107
  Change from Baseline at Week 12 (Primary Analysis in 2019) | -0.52 (6.193) | -0.56 (8.807)
  Change from Baseline at Week 24 (Primary Analysis in 2019): number analyzed (Participants) | 97 | 110
  Change from Baseline at Week 24 (Primary Analysis in 2019) | -0.65 (7.113) | -2.47 (8.833)
  Change from Baseline at Week 12 (Final Analysis in 2020): number analyzed (Participants) | 110 | 108
  Change from Baseline at Week 12 (Final Analysis in 2020) | -0.52 (6.193) | -0.89 (9.407)
  Change from Baseline at Week 24 (Final Analysis in 2020): number analyzed (Participants) | 97 | 111
  Change from Baseline at Week 24 (Final Analysis in 2020) | -0.65 (7.113) | -2.48 (8.893)
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.0874, rank ANCOVA — p-value was not adjusted for multiplicity and was provided for descriptive purpose only
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.1191, rank ANCOVA — p-values are not adjusted for multiplicity and are provided for descriptive purpose only

7. Secondary Outcome: Change in 6-minute Walk Distance (6MWD)
Description: Comparison of 6-minute walk distance before beginning and after completing study therapy.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter (m)
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
meter (m)
  Baseline | 391.6 (114.93) | 394.0 (108.09)
  Change from Baseline at Week 12: number analyzed (Participants) | 108 | 110
  Change from Baseline at Week 12 | -14.8 (66.23) | -7.7 (57.60)
  Change from Baseline at Week 24: number analyzed (Participants) | 99 | 108
  Change from Baseline at Week 24 | -2.0 (68.11) | -26.7 (79.32)
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.0395, rank ANCOVA — p-value was not adjusted for multiplicity and was provided for descriptive purpose only
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.0299, rank ANCOVA — p-value was not adjusted for multiplicity and was provided for descriptive purpose only

8. Secondary Outcome: Change in University of California, San Diego-Shortness of Breath Questionnaire Score
Description: University of California, San Diego Shortness of Breath Questionnaire (SOBQ) consists of 24-item on a scale of 0 to 5 with 0=not at all and 5=maximal or unable to do because of breathlessness. The total scores were calculated by summation of the 24 items scores and transformed into 0-100, with 0= poor quality of life , and 100= excellent quality of life.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Scores on a Scale
  Baseline: number analyzed (Participants) | 113 | 114
  Baseline | 44.17 (25.204) | 48.89 (23.441)
  Change from Baseline at Week 12: number analyzed (Participants) | 86 | 100
  Change from Baseline at Week 12 | 1.47 (19.707) | 2.24 (18.617)
  Change from Baseline at Week 24: number analyzed (Participants) | 84 | 102
  Change from Baseline at Week 24 | 5.21 (18.701) | 5.30 (22.078)
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.7788, rank ANCOVA; Analysis of Covariance Changes from baseline to week 24 are compared between the treatment arms using a rank ANCOVA; Hodges-Lehmann Median Difference = 0.00, 95% CI 2-sided [-5.00 to 5.00]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.8289, rank ANCOVA — Analysis of Covariance Changes from baseline to week 24 or early discontinuation visit are compared between the treatment arms using a rank ANCOVA with change from baseline as outcome variable and standardized rank baseline value as covariate; Hodges-Lehmann Median Difference = 0.00, 95% CI 2-sided [-5.00 to 5.00]

9. Secondary Outcome: Change in Score in Leicester Cough Questionnaire Score
Description: The Leicester Cough Questionnaire is a patient-reported questionnaire evaluating the impact of cough on quality of life. The questionnaire comprises 19 items. Each item assesses symptoms, or the impact of symptoms, over the last 2 weeks on a seven-point Likert scale. Scores in three domains (physical, psychological and social) were calculated as a mean for each domain (range 1 to 7). A total score (range 3 to 21) was also calculated by adding the domain scores together. Higher scores indicate better quality of life.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Scores on a Scale
  Baseline: number analyzed (Participants) | 127 | 125
  Baseline | 16.13 (3.711) | 15.15 (3.928)
  Change from Baseline at Week 12 (Primary Analysis in 2019): number analyzed (Participants) | 109 | 114
  Change from Baseline at Week 12 (Primary Analysis in 2019) | 0.35 (2.903) | -0.23 (3.654)
  Change from Baseline at Week 24 (Primary Analysis in 2019): number analyzed (Participants) | 100 | 114
  Change from Baseline at Week 24 (Primary Analysis in 2019) | 0.36 (2.889) | 0.04 (3.702)
  Change from Baseline at Week 12 (Final Analysis in 2020): number analyzed (Participants) | 109 | 114
  Change from Baseline at Week 12 (Final Analysis in 2020) | 0.35 (2.903) | -0.23 (3.654)
  Change from Baseline at Week 24 (Final Analysis in 2020): number analyzed (Participants) | 100 | 114
  Change from Baseline at Week 24 (Final Analysis in 2020) | 0.35 (2.884) | 0.04 (3.702)
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.1872, rank ANCOVA — p-value was not adjusted for multiplicity and was provided for descriptive purpose only; Analysis of Covariance Changes from baseline to week 24 are compared between the treatment arms using a rank ANCOVA; Hodges-Lehmann Median difference = 0.29, 95% CI 2-sided [-0.45 to 1.04]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.2019, rank ANCOVA — [p-value comment as in outcome 8, analysis 2]; Hodges-Lehmann Median Difference = 0.27, 95% CI 2-sided [-0.48 to 1.02]

10. Secondary Outcome: Change in Cough Visual Analog Scale (VAS) Score
Description: Cough VAS are 100-mm linear scales on which participants indicate the severity of their cough; 0 mm represents no cough and 100 mm the worst cough ever.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
millimeter (mm)
  Baseline: number analyzed (Participants) | 127 | 125
  Baseline | 35.60 (27.497) | 37.18 (26.270)
  Change from Baseline at Week 12: number analyzed (Participants) | 109 | 113
  Change from Baseline at Week 12 | -4.33 (20.017) | 3.32 (26.429)
  Change from Baseline at Week 24: number analyzed (Participants) | 100 | 114
  Change from Baseline at Week 24 | -2.52 (26.720) | 0.78 (30.121)
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.2995, rank ANCOVA; Analysis of Covariance Changes from baseline to week 24 are compared between the treatment arms using a rank ANCOVA; Hodges-Lehmann Median Difference = -2.00, 95% CI 2-sided [-10.00 to 4.00]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.3372, rank ANCOVA — [p-value comment as in outcome 8, analysis 2]; Hodges-Lehmann Median Difference = -2.00, 95% CI 2-sided [-10.00 to 4.00]

11. Secondary Outcome: Change in Total and Sub-scores of the Saint George's Respiratory Questionnaire (SGRQ)
Description: The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in participants with diseases of airways obstruction. Three component scores are: Symptoms (respiratory symptoms and severity); Activity (activities that cause or are limited by breathlessness); Impacts (social functioning and psychological disturbances due to airway disease). Each component sub-scores are calculated from the summed weights for the positive responses to questions. Total score summaries the impact of disease on overall health status. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status. It is calculated by summing all positive responses in the questionnaire and expressing the result as a percentage of the total weight for the questionnaire.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores of a Scale
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Scores of a Scale
  Symptoms sub-score - Baseline: number analyzed (Participants) | 126 | 125
  Symptoms sub-score - Baseline | 49.28 (21.687) | 53.10 (21.450)
  Change from Baseline in Symptoms sub-score at Week 12: number analyzed (Participants) | 107 | 114
  Change from Baseline in Symptoms sub-score at Week 12 | -2.60 (19.173) | 0.86 (16.212)
  Change from Baseline in Symptoms sub-score at Week 24: number analyzed (Participants) | 99 | 113
  Change from Baseline in Symptoms sub-score at Week 24 | -1.69 (19.186) | -0.66 (15.407)
  Activities sub-score - Baseline: number analyzed (Participants) | 123 | 123
  Activities sub-score - Baseline | 63.93 (20.388) | 66.96 (18.615)
  Change from Baseline in Activities sub-score at Week 12: number analyzed (Participants) | 106 | 112
  Change from Baseline in Activities sub-score at Week 12 | 1.17 (13.376) | 1.13 (13.704)
  Change from Baseline in Activities sub-score at Week 24: number analyzed (Participants) | 97 | 112
  Change from Baseline in Activities sub-score at Week 24 | 1.25 (14.629) | 2.22 (13.110)
  Impacts sub-score - Baseline: number analyzed (Participants) | 124 | 123
  Impacts sub-score - Baseline | 37.12 (20.484) | 41.47 (20.520)
  Change from Baseline in Impacts sub-score at Week 12: number analyzed (Participants) | 107 | 111
  Change from Baseline in Impacts sub-score at Week 12 | 0.29 (16.826) | 0.33 (13.888)
  Change from Baseline in Impacts sub-score at Week 24: number analyzed (Participants) | 97 | 112
  Change from Baseline in Impacts sub-score at Week 24 | -0.18 (13.884) | 1.07 (17.539)
  Total score - Baseline: number analyzed (Participants) | 123 | 123
  Total score - Baseline | 47.37 (18.465) | 51.46 (17.699)
  Change from Baseline in Total score at Week 12: number analyzed (Participants) | 106 | 112
  Change from Baseline in Total score at Week 12 | -0.17 (13.633) | 0.53 (11.724)
  Change from Baseline in Total score at Week 24: number analyzed (Participants) | 97 | 112
  Change from Baseline in Total score at Week 24 | 0.05 (12.549) | 0.85 (13.383)
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.1630, rank ANCOVA; Analysis of Covariance Changes from baseline to week 24 are compared between the treatment arms using a rank ANCOVA; Hodges-Lehmann Median Difference = -1.86, 95% CI 2-sided [-5.06 to 1.38]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.1851, rank ANCOVA — [p-value comment as in outcome 8, analysis 2]; Hodges-Lehmann Median Difference = -1.74, 95% CI 2-sided [-5.00 to 1.55]

12. Secondary Outcome: Number of Participants With Non-elective Hospitalization, Both Respiratory and All Cause
Description: Participants with non-elective hospitalization are reported.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 4
Measure: Number; unit: Number of Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Number of Participants
  All-cause hospitalization | 16 | 13
  Respiratory-related hospitalization | 5 | 5
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019. All-cause non-elective hospitalization; Test type: Superiority; p = 0.5922, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.59 to 2.49] — Hazard ratios and corresponding 95% CI are calculated by applying Cox-proportional hazard models
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019. Respiratory non-elective hospitalization; Test type: Superiority; p = 0.8057, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.26 to 2.83] — Hazard ratios and corresponding 95% CI are calculated by applying Cox-proportional hazard models
Statistical Analysis 3: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020. All-cause non-elective hospitalization; Test type: Superiority; p = 0.4613, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.63 to 2.73] — Hazard ratios and corresponding 95% CI are calculated by applying Cox-proportional hazard models
Statistical Analysis 4: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020. Respiratory non-elective hospitalization; Test type: Superiority; p = 0.9523, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.30 to 3.59] — Hazard ratios and corresponding 95% CI are calculated by applying Cox-proportional hazard models

13. Secondary Outcome: Percentage of Participants With Investigator-reported Acute Exacerbations
Description: Percentage of participants with acute exacerbation arereported.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Percentage of Participants | 3.9 | 5.6

14. Secondary Outcome: Time to First Investigator-reported Acute Exacerbations
Description: Time to first investigator reported acute exacerbations from start of treatment are reported.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Weeks | NA [NA to NA] — The end point could not be analyzed due to the limited number of events. | NA [NA to NA] — The end point could not be analyzed due to the limited number of events.
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Test type: Superiority; p = 0.7871, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.26 to 2.78]

15. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time to the first occurrence of a >10% absolute decline in percent predicted FVC, a >50 m decline of 6MWD, or death.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Week | 25.14 [24.14 to NA] — The end point could not be analyzed due to the limited number of events. | 24.71 [24.14 to NA] — The end point could not be analyzed due to the limited number of events.
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.3660, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.56 to 1.24]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.4173, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.57 to 1.26]

16. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time to the first occurrence of a >10% relative decline in percent predicted FVC, non-elective respiratory hospitalization, or death.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Week | NA [24.86 to NA] — The median was not reached in this analysis, thus an estimate cannot be calculated. In order to calculate the median time at least 50% of participants should report an event and this is not the case in this analysis due to low event number. | NA [24.14 to NA] — The median was not reached in this analysis, thus an estimate cannot be calculated. In order to calculate the median time at least 50% of participants should report an event and this is not the case in this analysis due to low event number.
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Primary Analysis in 2019; Test type: Superiority; p = 0.2726, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Cox Proportional Hazard = 0.79, 95% CI 2-sided [0.52 to 1.20]
Statistical Analysis 2: Comparison: Pirfenidone vs Placebo; Final Analysis in 2020; Test type: Superiority; p = 0.3386, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Cox Proportional Hazard = 0.82, 95% CI 2-sided [0.54 to 1.24]

17. Secondary Outcome: Time to Death From Any Cause
Description: Time to first documented death from start of treatment is reported.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Week | NA [NA to NA] — The end point could not be analyzed due to the limited number of events. | NA [NA to NA] — The end point could not be analyzed due to the limited number of events.
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Test type: Superiority; p = 0.9969, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms; Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.06 to 16.08]

18. Secondary Outcome: Time to Death From Respiratory Diseases
Description: Time to first documented death due to respiratory diseases from start of treatment will be reported.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 126
Week | NA [NA to NA] — The end point could not be analyzed due to the limited number of events. | NA [NA to NA] — The end point could not be analyzed due to the limited number of events.
Statistical Analysis 1: Comparison: Pirfenidone vs Placebo; Test type: Superiority; p = 0.3231, Log Rank; Log-rank tests based on the time to the first event are to compare the two treatment arms

19. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline (Day 1) to Week 28
Population: The safety population was defined as all participants with at least one intake of pirfenidone or placebo, i.e., at least one record in the drug-log of the double-blind period with a non-zero dose. Participants in the safety population were assigned to a treatment arm according to the actual treatment they received.
Measure: Number; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 124
Participants | 120 | 101

20. Secondary Outcome: Number of Participants With Dose Reductions and Treatment Interruptions During the Double-Blind Period
Description: Number of participants with dose reduction and treatment interruptions are reported.
Time Frame: From administration of the first dose of study drug to Week 24
Population: as for outcome 19
Measure: Number; unit: Number of Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 124
Number of Participants
  Participants with at least one dose modification | 51 | 34
  Participants with at least one dose interruption | 40 | 12

21. Secondary Outcome: Number of Participants With Dose Reductions and Treatment Interruptions During the 12-month Safety Follow-up
Description: Number of participants with dose reduction and treatment interruptions are reported.
Time Frame: From the Follow-up Visit at Week 28 through the follow-up period of 12 Months
Population: as for outcome 19
Measure: Number; unit: Number of Participants
Arm/Group | Open-Label Treatment (Pirfenidone) | Open-Label Treatment (Placebo)
Number analyzed (Participants) | 94 | 110
Number of Participants
  Participants with at least one dose modification | 41 | 60
  Participants with at least one dose interruption | 24 | 34

22. Secondary Outcome: Number of Participants Withdrawn From Trial Treatment or Trial Discontinuations During the Double-Blind Period
Description: Number of participants withdrawn from trial treatment or trial discontinuations are reported.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 19
Measure: Number; unit: Number of Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 127 | 124
Number of Participants | 25 | 12

23. Secondary Outcome: Number of Participants Withdrawn From Trial Treatment or Trial Discontinuations During the 12-month Safety Follow-up
Description: Number of participants withdrawn from trial treatment or trial discontinuations are reported.
Time Frame: From the Follow-up Visit at Week 28 through the follow-up period of 12 Months
Population: as for outcome 19
Measure: Number; unit: Number of Participants
Arm/Group | Open-Label Treatment (Pirfenidone) | Open-Label Treatment (Placebo)
Number analyzed (Participants) | 94 | 110
Number of Participants | 19 | 26

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to Week 28 in the double-blind period From the Follow-up Visit at Week 28 through the follow-up period of 12 Months in the open-label treatment period
Description: The safety population was defined as all participants with at least one intake of pirfenidone or placebo, i.e., at least one record in the drug-log of the double-blind period with a non-zero dose. Participants in the safety population were assigned to a treatment arm according to the actual treatment they received.
Arm/Group | Pirfenidone | Placebo | Open-Label Treatment (Pirfenidone) | Open-Label Treatment (Placebo)
All-Cause Mortality (participants affected / at risk) | 4/127 | 7/124 | 7/94 | 9/110
Serious Adverse Events (participants affected / at risk) | 18/127 | 20/124 | 26/94 | 27/110
Other Adverse Events (participants affected / at risk) | 107/127 | 81/124 | 64/94 | 86/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=127) | Placebo (N=124) | Open-Label Treatment (Pirfenidone) (N=94) | Open-Label Treatment (Placebo) (N=110)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung transplant rejection (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (6)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 6 (6)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (3) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 5 (7) | 3 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Polyp (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxocariasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=127) | Placebo (N=124) | Open-Label Treatment (Pirfenidone) (N=94) | Open-Label Treatment (Placebo) (N=110)
Constipation (Gastrointestinal disorders) | 7 (7) | 4 (4) | 6 (6) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 23 (27) | 23 (24) | 9 (16) | 15 (15)
Dyspepsia (Gastrointestinal disorders) | 17 (21) | 7 (7) | 5 (5) | 8 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 6 (7) | 7 (8) | 7 (7)
Nausea (Gastrointestinal disorders) | 40 (49) | 9 (10) | 15 (18) | 30 (39)
Vomiting (Gastrointestinal disorders) | 14 (17) | 6 (7) | 4 (6) | 18 (25)
Fatigue (General disorders) | 21 (22) | 19 (20) | 5 (5) | 12 (14)
Bronchitis (Infections and infestations) | 10 (11) | 3 (3) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 8 (10) | 13 (16) | 9 (12) | 14 (15)
Nasopharyngitis (Infections and infestations) | 7 (8) | 6 (9) | 10 (11) | 11 (11)
Respiratory tract infection (Infections and infestations) | 11 (11) | 5 (7) | 8 (9) | 9 (15)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 9 (10) | 10 (10) | 4 (5)
Weight decreased (Investigations) | 11 (11) | 6 (6) | 2 (2) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 18 (22) | 11 (11) | 7 (8) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 11 (13) | 13 (14) | 4 (4) | 8 (8)
Headache (Nervous system disorders) | 13 (19) | 4 (5) | 3 (3) | 12 (12)
Depression (Psychiatric disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 16 (17) | 10 (12) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 22 (25) | 9 (10) | 8 (8)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 8 (9) | 0 (0) | 2 (2) | 9 (12)
Rash (Skin and subcutaneous tissue disorders) | 9 (12) | 7 (8) | 8 (10) | 16 (19)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 10 (12)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 7 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT03099187/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03099187/SAP_003.pdf